CLINICAL TRIAL: NCT04013191
Title: An Open-Label, Parallel-Group, Pharmacokinetic, Safety and Tolerability Study of Single and Multiple Oral Administrations of Padsevonil in Adult and Elderly Study Participants
Brief Title: A Study to Test the Safety and Tolerability of Single and Multiple Doses of Padsevonil in Adult and Elderly Study Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UP0053
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Results first posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Elderly Study Participants; Adult Study Participants
Keywords: Padsevonil; Phase 1; Pharmacokinetic
MeSH Terms: interventions — padsevonil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adult study participants (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil
- Elderly study participants (Experimental): Participants will receive assigned single and multiple doses of padsevonil.
  Interventions: Drug: Padsevonil

INTERVENTIONS:
Drug: Padsevonil — Padsevonil will be administered in predefined dosages.

SUMMARY:
The purpose of the study is to evaluate the plasma pharmacokinetic of padsevonil in adult and elderly study participants.

ELIGIBILITY:
Inclusion Criteria:

* Study participants in the adult cohort must be ≥18 to 64 years of age at the time of signing the informed consent form (ICF)
* Study participants in the elderly cohort must be ≥65 years of age at the time of signing the ICF
* Study participants who are overtly healthy as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring. In addition, elderly study participants must be considered to be in general good physical and mental health
* Study participants must have a body weight of at least 50 kg for males and 45 kg for females, and a body mass index within the range of 18 to 32 kg/m2 (inclusive)

Exclusion Criteria:

* Study participant has a current or past psychiatric condition that, in the opinion of the Investigator, could compromise the study participant's safety or ability to participate in this study, or a history of schizophrenia or other psychotic disorder, bipolar disorder, or severe unipolar depression. The presence of potential psychiatric exclusion criteria will be determined based on the psychiatric history collected at Screening
* Study participant has history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data
* Study participant has a known hypersensitivity to any components of the study medication as stated in this protocol
* Subject has a history of unexplained syncope or a family history of sudden death due to long QT syndrome
* Study participant has abnormal blood pressure
* Study participant has had lymphoma, leukemia, or any malignancy within the past 5 years, except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Study participant has a lifetime history of suicide attempt, or has had suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the "Screening/Baseline" version of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening
* Study participant has past or intended use of over-the-counter or prescription medication, including herbal medications within 2 weeks or 5 half-lives prior to dosing
* The study participant has used hepatic enzyme-inducing drugs within 2 months prior to dosing
* Study participant has previously received padsevonil (PSL) in this or another study
* Study participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN)
* Study participant has bilirubin >1.0xULN (isolated bilirubin >1.0xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Study participant has current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Study participant has any clinically relevant electrocardiogram (ECG) finding at Screening or at Baseline. Study participant has an abnormality in the 12-lead ECG that, in the opinion of the Investigator, increases the risks associated with participating in the study. In addition, any study participant with any of the following findings will be excluded: (a) QT interval corrected for heart rate using Bazett's formula (QTcB) or Fridericia's formula (QTcF) >450 ms in study participants in 2 of 3 ECG recordings; (b) other conduction abnormalities (defined as PR interval ≥220 ms); (c) irregular rhythms other than sinus arrhythmia or occasional, rare supraventricular or rare ventricular ectopic beats. In case of an out of range result, 1 repeat will be allowed. If out of range again, the study participant cannot be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (1):
- Up0053 001, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, Individual Patient Data cannot be adequately anonymized and there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll patients in July 2019 and concluded in October 2019.
Pre-assignment Details: The study included a 28 days Screening period, a 21 days Treatment period: Period 1A single dose (SD) on Days 1 to 7 and Period 1B multiple dose (MD) on Days 8 to 21 and a Safety Follow-up period on Day 22.
  Participant Flow refers to the Full Analysis Set.
Groups:
- Adults (18-64 Years); Elderly (>= 65 Years): Participants received assigned single and multiple doses of padsevonil.
Period: Overall Study
Arm/Group | Adults (18-64 Years) | Elderly (>= 65 Years)
Started | 10 | 18
Completed Period 1A (Single Dose) | 10 | 18
Completed Period 1B (Multiple Dose) | 9 | 18
Completed | 9 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to Full Analysis Set (FAS) which consisted of all study participants who signed the informed consent form (ICF) and received at least 1 dose of PSL.
Arm/Group | Adults (18-64 Years) | Elderly (>= 65 Years) | Total Title
Number analyzed (Participants) | 10 | 18 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 10
  >=65 years | 0 | 18 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.2) | 69.7 (4.5) | 60.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 4 | 9 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 0 | 1
  White | 9 | 18 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Maximum Plasma Concentration (Cmax) of a Single Dose Padsevonil (PSL)
Description: Cmax was measured in nanograms per milliliter (ng/mL).
Time Frame: Plasma samples were taken predose on Day 1 and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose
Population: The Pharmacokinetic-Per Protocol Set (PK-PPS) was a subset of the FAS, consisting of study participants who had no important protocol deviation (IPD) affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Adults (18-64 Years) (PK-PPS): Participants received assigned single and multiple doses of padsevonil, forming the Pharmacokinetic-Per Protocol Set (PK-PPS).
- Elderly (>= 65 Years) (PK-PPS): Participants received assigned single and multiple doses of padsevonil, forming the PK-PPS.
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 10 | 18
ng/mL | 903.6 [712 to 1150] | 838.4 [702 to 1000]
Statistical Analysis 1: Comparison: Adults (18-64 Years) (PK-PPS) vs Elderly (>= 65 Years) (PK-PPS); The analysis of variance (ANOVA) model included the fixed effects of age group. The natural logs were taken of the dependent variables and back-transformed after the analysis; Test type: Other; ANOVA; Point Estimate = 0.928, 90% CI 2-sided [0.725 to 1.19]

2. Primary Outcome: The Area Under the Curve From 0 to t (AUC0-t) of a Single Dose Padsevonil (PSL)
Description: AUC0-t: area under the plasma concentration-time curve from time 0 to the last quantifiable concentration. It was measured in hours times nanograms per milliliter (h*ng/mL).
Time Frame: Plasma samples were taken predose on Day 1 and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 10 | 18
h*ng/mL | 4915 [3630 to 6650] | 6011 [4800 to 7530]
Statistical Analysis 1: Comparison: Adults (18-64 Years) (PK-PPS) vs Elderly (>= 65 Years) (PK-PPS); The ANOVA model included the fixed effects of age group. The natural logs were taken of the dependent variables and back-transformed after the analysis; Test type: Other; ANOVA; Point Estimate = 1.22, 90% CI 2-sided [0.894 to 1.67]

3. Primary Outcome: The Area Under the Curve (AUC) of a Single Dose Padsevonil (PSL)
Description: AUC was measured in hours times nanograms per milliliter (h*ng/mL).
Time Frame: Plasma samples were taken predose on Day 1 and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8, 12, 24, 48 and 72 hours postdose
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 10 | 18
h*ng/mL | 4950 [3650 to 6720] | 6061 [4830 to 7610]
Statistical Analysis 1: Comparison: Adults (18-64 Years) (PK-PPS) vs Elderly (>= 65 Years) (PK-PPS); [analysis description as in outcome 2, analysis 1]; Test type: Other; ANOVA; Point Estimate = 1.22, 90% CI 2-sided [0.893 to 1.68]

4. Primary Outcome: The Maximum Plasma Concentration at Steady-state (Cmax, ss) of Multiple Doses Padsevonil (PSL)
Description: Cmax, ss was measured in nanograms per milliliter (ng/mL).
Time Frame: Plasma samples were taken predose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 12 hours on Day 13
Population: The PK-PPS was a subset of the FAS, consisting of study participants who had no IPD affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter. 1 participant in the adult cohort discontinued due to a treatment emergent adverse event (TEAE) after 5 days of PSL administration in the MD Period.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 9 | 18
ng/mL | 1157 [942 to 1420] | 1180 [1020 to 1360]
Statistical Analysis 1: Comparison: Adults (18-64 Years) (PK-PPS) vs Elderly (>= 65 Years) (PK-PPS); [analysis description as in outcome 2, analysis 1]; Test type: Other; ANOVA; Point Estimate = 1.02, 90% CI 2-sided [0.829 to 1.26]

5. Primary Outcome: The Area Under the Curve (AUCtau) Over a Dosing Interval of Multiple Doses Padsevonil (PSL)
Description: AUCtau was measured in hours times nanograms per milliliter (h*ng/mL).
Time Frame: Plasma samples were taken predose and 0.25, 0.5, 0.75, 1, 1.5, 3, 4, 6, 8 and 12 hours on Day 13
Population: The PK-PPS was a subset of the FAS, consisting of study participants who had no IPD affecting the PK parameters and for whom a sufficient number of samples were available to determine at least 1 PK parameter. 1 participant in the adult cohort discontinued due to a TEAE after 5 days of PSL administration in the MD Period.
Measure: Least Squares Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 9 | 18
h*ng/mL | 5346 [4130 to 6920] | 6307 [5260 to 7570]
Statistical Analysis 1: Comparison: Adults (18-64 Years) (PK-PPS) vs Elderly (>= 65 Years) (PK-PPS); [analysis description as in outcome 2, analysis 1]; Test type: Other; ANOVA; Point Estimate = 1.18, 90% CI 2-sided [0.908 to 1.53]

6. Secondary Outcome: The Amount of Padsevonil (PSL) Excreted in Urine
Description: Samples were taken to assess the amount of padsevonil that was excreted in urine. Ae,ss refers to cumulative amount of PSL excreted in the urine at steady state.
Time Frame: Urine samples were taken on Day 1, Day 2, Day 3, Day 4 and Day 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 10 | 18
milligrams
  Single dose: Day 1 (Ae) | 0.0862 (153.9) | 0.0979 (45.9)
  Multiple dose: Day 13 (Ae,ss): number analyzed (Participants) | 9 | 18
  Multiple dose: Day 13 (Ae,ss) | 0.0924 (109.5) | 0.166 (45.5)
  Metabolite 1, Single dose: Day 1 (Ae) | 0.941 (79.9) | 1.13 (20.3)
  Metabolite 1, Multiple dose: Day 13 (Ae,ss): number analyzed (Participants) | 9 | 18
  Metabolite 1, Multiple dose: Day 13 (Ae,ss) | 1.16 (96.9) | 1.86 (35.9)
  Metabolite 2, Single dose: Day 1 (Ae) | 18.7 (68.3) | 14.6 (54.2)
  Metabolite 2, Multiple dose: Day 13 (Ae,ss): number analyzed (Participants) | 9 | 18
  Metabolite 2, Multiple dose: Day 13 (Ae,ss) | 13.3 (79.5) | 14.4 (45.9)

7. Secondary Outcome: The Ratio of Padsevonil (PSL) to Its Metabolites Excreted in Urine
Description: Samples were taken to assess the metabolic ratio of padsevonil that was excreted in urine. MRAe was defined as the metabolic ratio of PSL to its metabolites for cumulative amount of PSL metabolites excreted in the urine. ss refers to steady state.
Time Frame: Urine samples were taken on Day 1, Day 2, Day 3, Day 4 and Day 13
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Adults (18-64 Years) (PK-PPS) | Elderly (>= 65 Years) (PK-PPS)
Number analyzed (Participants) | 10 | 18
ratio
  Metabolite 1, Single dose: Day 1 (MRAe) | 10.6 (52.8) | 11.2 (40.3)
  Metabolite 1, Multiple dose: Day 13 (MRAe,ss): number analyzed (Participants) | 9 | 18
  Metabolite 1, Multiple dose: Day 13 (MRAe,ss) | 12.2 (43.9) | 10.9 (38.2)
  Metabolite 2, Single dose: Day 1 (MRAe) | 217 (122.3) | 149 (81.8)
  Metabolite 2, Multiple dose: Day 13 (MRAe,ss): number analyzed (Participants) | 9 | 18
  Metabolite 2, Multiple dose: Day 13 (MRAe,ss) | 144 (81.1) | 86.8 (67.7)

8. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. An AE could, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study medication.
Time Frame: From Baseline until End-of-Treatment visit (up to Day 22)
Population: The Full Analysis Set (FAS) consisted of all study participants who signed the informed consent form (ICF) and received at least 1 dose of PSL.
Measure: Count of Participants; unit: Participants
Groups:
- Adults (18-64 Years) (FAS): Participants received assigned single and multiple doses of padsevonil, forming the Full Analysis Set (FAS).
- Elderly (>= 65 Years) (FAS): Participants received assigned single and multiple doses of padsevonil, forming the FAS.
Arm/Group | Adults (18-64 Years) (FAS) | Elderly (>= 65 Years) (FAS)
Number analyzed (Participants) | 10 | 18
Participants
  Single Dose Period (1A) | 10 | 18
  Multiple Dose Period (1B) | 10 | 17

9. Secondary Outcome: Number of Participants With Serious Adverse Events
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  * Results in death
  * Is life-threatening
  * Requires in patient hospitalization or prolongation of existing hospitalization
  * Is a congenital anomaly or birth defect
  * Is an infection that requires treatment parenteral antibiotics
  * Other important medical events which based on medical or scientific judgement may jeopardize the patients, or may require medical or surgical intervention to prevent any of the above
Time Frame: From Baseline until End-of-Treatment visit (up to Day 22)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Adults (18-64 Years) (FAS) | Elderly (>= 65 Years) (FAS)
Number analyzed (Participants) | 10 | 18
Participants
  Single Dose Period (1A) | 0 | 0
  Multiple Dose Period (1B) | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Leading to Discontinuation of the Study
Description: An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Baseline until End-of-Treatment visit (up to Day 22)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Adults (18-64 Years) (FAS) | Elderly (>= 65 Years) (FAS)
Number analyzed (Participants) | 10 | 18
Participants
  Single Dose Period (1A) | 0 | 0
  Multiple Dose Period (1B) | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Baseline until End-of-Treatment visit (up to Day 22)
Groups:
- Adults (18-64 Years) (FAS) SD Period (1A); Elderly (>= 65 Years) (FAS) SD Period (1A): Participants received a single dose of padsevonil during Period (1A), forming the FAS.
- Adults (18-64 Years) (FAS) MD Period (1B); Elderly (>= 65 Years) (FAS) MD Period (1B): Participants received multiple doses of padsevonil during Period (1B), forming the FAS.
Arm/Group | Adults (18-64 Years) (FAS) SD Period (1A) | Elderly (>= 65 Years) (FAS) SD Period (1A) | Adults (18-64 Years) (FAS) MD Period (1B) | Elderly (>= 65 Years) (FAS) MD Period (1B)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/18 | 0/10 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/18 | 0/10 | 0/18
Other Adverse Events (participants affected / at risk) | 10/10 | 18/18 | 10/10 | 17/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adults (18-64 Years) (FAS) SD Period (1A) (N=10) | Elderly (>= 65 Years) (FAS) SD Period (1A) (N=18) | Adults (18-64 Years) (FAS) MD Period (1B) (N=10) | Elderly (>= 65 Years) (FAS) MD Period (1B) (N=18)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 9 (9) | 17 (17) | 10 (10) | 16 (16)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 4 (4) | 6 (6)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disinhibition (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enuresis (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT04013191/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/91/NCT04013191/SAP_001.pdf